CLINICAL TRIAL: NCT03011489
Title: Parent's Satisfaction and Evaluation of Postsurgical Outcomes in Unilateral Cleft Lip / Palate Newly Born Infants With / Without Vacuum Formed Nasoalveolar Molding Aligners : A Controlled Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Khadega Ali Al Khateeb, Master student, faculty of oral and dental medicine, Cairo university, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UCLP_Vacuum
Record Dates: First submitted 2017-01-04; First posted 2017-01-05 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Cleft Lip and Palate
MeSH Terms: conditions — Cleft Lip

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vacuum formed aligners group (Experimental): This group will receive Vacuum formed aligners in addition to taping for 3 Months with follow-up every 1-2 weeks
  Interventions: Device: Vacuum formed aligners
- control group (No Intervention): This group will not receive any treatment

INTERVENTIONS:
Device: Vacuum formed aligners — Infants will receive this appliance which is a maxillary plate with nasal stent in addition to taping on the upper lip (taping is a modified step in Figueroa's technique.
  Arms: Vacuum formed aligners group

SUMMARY:
Newborns with unilateral cleft lip/ palate will be treated pre-surgically by Vacuum formed aligners in order to evaluate its effect on Nasoalveolar complex.

DETAILED DESCRIPTION:
newborns with unilateral cleft lip/ palate will be allocated into two groups: treatment group will receive Vacuum formed aligners while control group will not receive Vacuum formed aligners.

the follow-up period will be 3 months till surgical lip closure. the assessment will be through a questionnaire for the parents' satisfaction outcome, standardized photographs for measurement of nasal changes and interlabial gap outcome and digital maxillary models for the maxillary dimension change outcome.

ELIGIBILITY:
Inclusion Criteria:

* Non-syndromic Infants with complete unilateral cleft lip and palate
* Infants less than 3 months of age
* Males and females.
* Infants with displaced alveolus
* Patients whose parents provided written consent for the study.

Exclusion Criteria:

* Patients above 3 months of age
* Syndromic, malnourished and systemically ill infants.
* Patients with bilateral cleft lip and palate.
* Incomplete Cleft lip.
* Medically compromised patients
* Patient's/guardians who will be unwilling to go through the PNAM therapy

Ages: 1 Week to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 14 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Parents' satisfaction | 3 months
  It will be measured by questionnaire

SECONDARY OUTCOMES:
Changes in Nasal morphology( Height, width, angulation of columella | 3 months
  It will be measured in mm by Standardized Digital photographs
Changes in Interlabial gab | 3 months
  It will be measured in mm by Standardized Digital photographs
Changes in Maxillary arch dimension | 3 months
  It will be measured in mm by Digital models

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Abdu Abdelsayed, professor, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: No